CLINICAL TRIAL: NCT04514211
Title: The Effects of Propofol and Sevoflurane on Postoperative Heart Rate Variability and Postoperative Nausea Vomiting
Brief Title: Heart Rate Variability and Postoperative Nausea Vomiting
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, assistant professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-20-293
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting; heart rate variability; propofol; sevoflurane
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol: General anesthesia using propofol infusion
  Interventions: Drug: Propofol
- Sevoflurane: General anesthesia using sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — General anesthesia using propofol infusion
  Other Names: Propofol infusion
  Groups: Propofol
Drug: Sevoflurane — General anesthesia using sevoflurane
  Other Names: Sevoflurane inhalation
  Groups: Sevoflurane

SUMMARY:
Propofol and sevoflurane have different effects on heart rate variability. It has not yet been reported whether this difference in effect remains at recovery time after anesthesia and the difference is related to postoperative nausea and vomiting has not been studied. The aim of this study is observe whether propofol and sevoflurane have different effects on heart rate variability during recovery and the differences can predict the occurrence of postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Different types of anesthetics have different effects on heart rate variability. However It has not yet been reported whether this difference in effect remains at recovery time after anesthesia.

Several studies have been reported that preoperative heart rate variability predicted the occurence of postoperative nausea and vomiting. However, whether the difference in heart rate variability after anesthesia is related to the difference in postoperative nausea and vomiting has not been studied. Therefore, this study aims to observe whether propofol and sevoflurane have differences during recovery period after anesthesia in heart rate variabiliy. In addition, we want to examine that these differences during recovery period in heart rate variability can predict the occurrence of nausea and vomiting within 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled breast surgery under general anesthesia

Exclusion Criteria:

* Arrhythmia
* Uncooperative with the measuring heart rate variability
* Diabetes
* Hypertension on medication
* Patients taking psychiatric drugs
* Thyroid disease

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Include only mathces self-representation of gender identity and biological sex
Study Population: 20~50 years old female patients who scheduled breast surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
heart rate variability in recovery room | within 1 hour
  Postoperative heart rate variability measuring at recovery room Frequency domain result: total power, low frequency power, high frequency power, Low frequency/high frequency power ratio

SECONDARY OUTCOMES:
Postoperative nausea vomiting impact scale | 48 hours after anesthesia
  Q1. Have you vomited or had dry-retching? 0. No
  1. Once
  2. twice
  3. 3 or more times
  Q2. Have you experienced a feeling of nausea? If yes, has your feeling of nausea interfered with activities of daily living? 0. not at all
  1. Sometimes
  2. often or most of the time
  3. All of the time
  Add the numerical responses to questions 1 and 2. (total score 0~6)
The incidence of postoperative nausea and vomiting | 48 hours after anesthesia
  the time of occurence
Patient's satisfaction about postoperative nausea and vomiting | 48 hours after anesthesia
  verbal rating scale (0~10), 0=very unsatisfied, 10=very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We will provide it upon the reasonable personal request.